CLINICAL TRIAL: NCT03620851
Title: Effect of Age on the Efficiency of Enhanced Recovery Program After Colorectal Surgery
Brief Title: Enhanced Recovery Program After Colorectal Surgery in Elderly (ERPOLD)
Acronym: ERPOLD
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor in Anesthesiology, University of Liege
Other Study IDs: ERPELDERLY
Record Dates: First submitted 2018-07-18; First posted 2018-08-08 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Surgery
Keywords: enhanced recovery program; colorectal surgery; elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly patients (≥70 yo) vs. younger patients (<70 yo): elderly patients (≥ 70 yo) and younger patients (< 70 yo)
  Interventions: Other: effect of age

INTERVENTIONS:
Other: effect of age — effect of age on the efficiency of enhanced recovery program

SUMMARY:
Comparison of the efficiency of enhanced recovery program after colorectal surgery in elderly patients (≥ 70 yo) and younger patients (< 70 yo). Efficiency will be rated as a function of length of hospital stay, postoperative complications (medical and surgical, as well as adherence to protocol.

DETAILED DESCRIPTION:
In 1995 Henrik Kehlet described the concept of fast track surgery after colectomy. It consisted of a multimodal and multidisciplinary approach that aimed at controlling the surgical stress response and at mitigating its consequences. Subsequently postoperative recovery is improved and accelerated, which allows a median hospital stay of 2-days after laparoscopic colectomy. The concept of fast track surgery progressively evolved into enhanced recovery programme (ERP). The acceleration of postoperative recovery and the reduction in the duration of hospitalisation are not associated with an increased incidence of surgical complications nor a greater rate of unplanned hospital readmission, but rather result in less medical complications. The economic benefits are obvious.

The elderly present specific physical, metabolic and socio-environmental characteristics that should be considered in case of surgery. Age has been shown to be an independent prognostic factor for postoperative morbidity after colorectal surgery, but this was reported before the development of ERP. Indeed implementation of ERP significantly reduces the rate of postoperative complications, even in the elderly. Increased risk of postoperative morbidity in elderly as compared to younger patients is nevertheless commonly admitted. Moreover adherence of elderly with the items of ERP is usually considered inferior than that of younger patients. Adaptation of ERP to the specificities of elderly is sometimes advocated. All these explain the reluctance of many practitioners to propose ERP in older patients. However recent meta-analyses suggest that implementation of ERP is feasible and efficient in these patients. The retrospective analysis of our first 100 patients introduced in our audit database revealed even similar length of hospital stay for elderly and younger patients.

The investigators therefore compared the length of hospital stay in the elderly and the younger patients and tested the hypothesis of non-inferiority for elderly patients as compared to younger patients. This is a retrospective analysis of 270 consecutive patients scheduled for colorectal surgery, all managed with the same ERP protocol, and prospectively introduced in our audit database.

ELIGIBILITY:
Inclusion Criteria:

• All patients scheduled for colorectal surgery since November 2015

Exclusion Criteria:

• Emergency surgery

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients scheduled for colorectal surgery have been included in an enhanced recovery program (ERP) since the 1st November 2015. Preoperative characteristics, surgical and anesthetic data, as well postoperative parameters and complications have been entered prospectively in the GRACE (Groupe francophone de Réhabilitataion Améliorée après ChirurgiE)
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
length of hospital stay after colorectal surgery (day) | through study completion, an average of 1 month
  The duration of hospitalization is defined as the numberof days the patient stays in the hospital between the day of his surgery and the day of his discharge from the hospital

SECONDARY OUTCOMES:
postoperative complications after colorectal surgery | through study completion, an average of 1 month
  The incidence of postoperative complications (medical and surgical) occurring during the hospital stay and up-to 30-day after surgery will be recorded from our audit database. The following medical complications will be recorded: cardiac, pulmonary, neurological, and uro-nephrologic complications. For surgical complications, we will record postoperative ileus, parietal complications, anastomotic leakage, intra-abdominal sepsis and hemorrhage, unplanned surgery.
adherence to the enhanced recovery program | through study completion, an average of 1 month
  compliance to the different items of the program

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Joris, MD, Principal Investigator — CHU Liege, Belgium
Locations (1):
- CHU Liége, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joris J, Hans G, Coimbra C, Decker E, Kaba A. Elderly patients over 70 years benefit from enhanced recovery programme after colorectal surgery as much as younger patients. J Visc Surg. 2020 Feb;157(1):23-31. doi: 10.1016/j.jviscsurg.2019.07.011. Epub 2019 Jul 31. PMID 31377111